CLINICAL TRIAL: NCT00479739
Title: Randomised, Double-blind, Double-dummy, 52-week, Parallel Group Study of a Standard Dosing Regimen With Salmeterol/Fluticasone propionate50/250 Twice Daily Diskus Versus a Symptom-driven, Variable Dosing Regimen With Formoterol/Budesonide Combination 4.5/160 in Adult Asthmatics
Brief Title: CONCEPT: A 1-Year Comparison Of A Stable Dose Of SERETIDE® Inhaler With An Adjustable Maintenance Dose Of SYMBICORT® Inhaler. SERETIDE® Inhaler is a Trademark of GSK Group of Companies. SYMBICORT® Inhaler is a Trademark of Astra Zeneca.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM40056
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: formoterol/budesonide; exacerbations; Salmeterol/fluticasone propionate; adjustable maintenance dosing; asthma control
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Salmeterol/fluticasone propionate or formoterol/budesonide

INTERVENTIONS:
Drug: Salmeterol/fluticasone propionate or formoterol/budesonide

SUMMARY:
To compare a stable dose of salmeterol/fluticasone propionate with a variable dose of formoterol/budesonide where the dose is adjusted according to a physician-guided self-management plan

DETAILED DESCRIPTION:
A randomised, double-blind, double-dummy, 52-week, parallel group study of a standard dosing regimen with salmeterol/fluticasone propionate combination 50/250mcg bid (via the DISKUS/ACCUHALER inhaler) versus a symptom-driven variable dosing regimen with formoterol/budesonide combination 6/200mcg (via a breath-actuated dry powder reservoir inhaler)in adults asthmatics

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history of asthma
* Forced expiratory volume in 1 second between 60% and 90% of predicted
* Using an inhaled corticosteroid (ICS)at a dose equivalent to 200 to 500 mcg daily of beclomethasone (BDP)or equivalent combined with a long-acting beta-2-agonist or an ICS alone at a dose equivalent to >500 to 1000mcg daily of BDP daily

Exclusion Criteria:

* Lower respiratory tract infection within 1 month of study entry
* Use of systemic corticosteroids within 1 month of study entry
* Smoking history of 10 pack years or more Changes in regular asthma therapy within 12 weeks of study entry
* Any significant disorder that in the investigator's opinion might put the patient at risk or influence the study outcomes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2002-11; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Mean percentage of symptom-free days over a 52-week treatment period

SECONDARY OUTCOMES:
Mean percentage of rescue-free days Daily asthma symptom scores Daily rescue usage Mean morning peak flow Percentage of nights awoken due to asthma Rate of exacerbations Airway hyper-responsiveness(PC20 AMP)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (86):
- Australia (4):
  - GSK Investigational Site, Balmain, New South Wales
  - GSK Investigational Site, Brisbane, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Toorak Gardens, South Australia
- Austria (2):
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Vienna
- Belgium (8):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Ath
  - GSK Investigational Site, Gilly
  - GSK Investigational Site, Hornu
  - GSK Investigational Site, Leopoldsburg
  - GSK Investigational Site, Oostham
  - GSK Investigational Site, Tessenderlo
  - GSK Investigational Site, Tienen
- Bulgaria (4):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (11):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Maple Ridge, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- Estonia (3):
  - GSK Investigational Site, Kohtal-Jdrve
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (6):
  - GSK Investigational Site, Jakobstad
  - GSK Investigational Site, Joensuu
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Raahe
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Varkaus
- Germany (7):
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Lahr, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Berlin, State of Berlin
- Ireland (6):
  - GSK Investigational Site, Blackpool, Cork
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
  - GSK Investigational Site, Kilkenny
  - GSK Investigational Site, Lifford
  - GSK Investigational Site, Tallaght, Dublin
- Latvia (3):
  - GSK Investigational Site, Limbaži
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Valmiera
- Netherlands (13):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Bennebroek
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Geldermalsen
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Losser
  - GSK Investigational Site, Made
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Spijkenisse
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Voerendaal
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch Hospital
- GSK Investigational Site, Skopje, North Macedonia
- Spain (9):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Las Palmas
  - GSK Investigational Site, Lugo
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Valencia
- United Kingdom (7):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Saffron Walden, Essex
  - GSK Investigational Site, Barry, Glamorgan
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Fleetwood

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Boulet LP, Fitzgerald M, Pieters R. The CONCEPT study: comparative influence of two treatment strategies on airway response to AMP. European Respiratory Journal Supplement 2005; 26: 429.
- [Result] FitzGerald JM, Boulet LP, Follows RM. The CONCEPT trial: a 1-year, multicenter, randomized,double-blind, double-dummy comparison of a stable dosing regimen of salmeterol/fluticasone propionate with an adjustable maintenance dosing regimen of formoterol/budesonide in adults with persistent asthma. Clin Ther. 2005 Apr;27(4):393-406. doi: 10.1016/j.clinthera.2005.03.006. PMID 15922813
- [Result] Fitzgerald M, Boulet LP, Pieters WR. Improved control of symptoms and exacerbations with stable dose treatment with salmeterol/fluticasone propionate compared with adjustable maintenance dosing with formoterol/budesonide. European Respiratory Journal Supplement 2005; 26: 429.
- [Result] Price D, Williams AE, Yoxall S. Quality of life of stable dose treatment with salmeterol/fluticasone compared with adjustable maintenance dosing with formoterol/budesonide. European Respiratory Journal Supplement 2005; 26(Suppl. 49): 252 (plus poster) abstr. P1720.
- [Derived] Price DB, Williams AE, Yoxall S. Salmeterol/fluticasone stable-dose treatment compared with formoterol/budesonide adjustable maintenance dosing: impact on health-related quality of life. Respir Res. 2007 Jul 4;8(1):46. doi: 10.1186/1465-9921-8-46. PMID 17610727
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: SAM40056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAM40056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAM40056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAM40056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAM40056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAM40056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAM40056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register